CLINICAL TRIAL: NCT03018223
Title: A Calcineurin Inhibitor-Free GVHD Prevention Regimen After Related Haploidentical Peripheral Blood Stem Cell Transplantation
Brief Title: Calcineurin Inhibitor-Free GVHD Prevention Regimen After Related Haplo PBSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18766
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Non-Hodgkin's Lymphoma; Acute Leukemia in Remission; Chronic Myeloid Leukemia; Primary Myelofibrosis; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Hodgkin Lymphoma; Multiple Myeloma
Keywords: Acute leukemia in CR; Chronic myeloid leukemia; Non-Hodgkin lymphoma in high risk; Graft vs. Host Disease; GVHD; Hematopoietic cell transplant (HCT)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Hodgkin Disease; Multiple Myeloma; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Busulfan; Cyclophosphamide; Whole-Body Irradiation; Radiotherapy; Sirolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Conditioning/HCT/GVHD Prophylaxis (Experimental): Pre-HCT Conditioning, HCT, GVHD Prophylaxis.
  1. Conditioning regimen: To reduce heterogeneity, two commonly used myeloablative (MAC) and reduced intensity (RIC) regimens are permitted on this trial. Myeloablative conditioning: fludarabine, busulfan. Reduced intensity conditioning: fludarabine, cyclophosphamide, total body irradiation.
  2. Peripheral blood hematopoietic cell transplantation
  3. Graft vs. Host Disease (GVHD) prevention treatment: cyclophosphamide, mycophenolate mofetil, sirolimus.
  4. Growth factor support: G-CSF
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Cyclophosphamide; Radiation: Total body irradiation (TBI); Procedure: Peripheral Blood Hematopoietic Cell Transplantation (HCT); Drug: Sirolimus (SIR); Drug: Mycophenolate mofetil (MMF); Drug: Granulocyte-colony stimulating factor (G-CSF)

INTERVENTIONS:
Drug: Fludarabine — Myeloablative conditioning: 40 mg/m^2 daily for 4 days. Dose will be adjusted for estimated creatinine clearance. Reduced intensity conditioning: 30 mg/m^2 daily on days -6, -5, -4, -3 and -2. Dose will be adjusted for estimated creatinine clearance.
  Other Names: Fludara, Oforta
Drug: Busulfan — Myeloablative conditioning: IV dosing targeted for a daily total area under curve (AUC) 5300 mmol*min/L for 4 days. Busulfan AUC will be pharmacokinetically targeted. An AUC 3500 mmol*min/l may be considered in patients over 60 years of age or with multiple comorbidities. Chemotherapy may start on day -6 or day -5 depending on the day of admission (-6 for Wednesday admission, -5 for Sunday admission).
  Other Names: Busulfex, Myleran
Drug: Cyclophosphamide — Reduced intensity conditioning: 14.5 mg/kg/day on days -6, -5. GVHD prophylaxis: 50 mg/kg ideal body weight (IBW) daily dose will be given on days +3 and +4 post-transplant as an IV infusion over 1-2 hours.
  Other Names: Cytoxan
Radiation: Total body irradiation (TBI) — Reduced intensity conditioning: 200 centigray (cGy) on day -1.
  Other Names: radiotherapy
Procedure: Peripheral Blood Hematopoietic Cell Transplantation (HCT) — On day 0, patients will receive a peripheral blood hematopoietic cell graft.
  Other Names: cell graft
Drug: Sirolimus (SIR) — GVHD prophylaxis: SIR will be administered as a 9 mg oral loading dose on day +5, followed by maintenance. SIR levels will be monitored and maintenance dosing adjusted as needed for a target trough level 8 to 14 ng/ml, per Moffitt BMT program standard practice. In the absence of acute GVHD, sirolimus taper will start on day +90 (+/- 10 days) and it is suggested to finish by day +180.
  Other Names: Rapamune
Drug: Mycophenolate mofetil (MMF) — GVHD prophylaxis: MMF will start on day +5 at a dose of 15 mg/kg every 8 hours IV with the maximum daily dose not to exceed 3 gm. MMF will be changed to orally (PO) and discontinued on day +35 (without taper) in the absence of acute GVHD.
  Other Names: CellCept
Drug: Granulocyte-colony stimulating factor (G-CSF) — Growth factor support: G-CSF will be given beginning on day 5 at a dose of 5 mcg/kg/day (rounding to the nearest vial dose), until absolute granulocyte count (ANC) is > 1,000/mm^3 for three consecutive days. G-CSF may be given IV or subcutaneously.
  Other Names: Neupogen, Filgrastim

SUMMARY:
The purpose of this study is to find out if a combination of drugs (these are called: cyclophosphamide, sirolimus, and mycophenolate mofetil) will protect participants better against graft vs. host disease (GVHD) after receiving a hematopoietic cell transplant from a related partially matched (haploidentical) donor. As part of the treatment for their blood cancer, participants need a hematopoietic cell transplantation (HCT) to improve their chances of cure. In any HCT, after the stem cell infusion is given, a combination of drugs is needed to prevent GVHD and facilitate acceptance of the graft.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants:

* Age: Must be older than 18 years, no upper age limit.
* Karnofsky performance status: Full intensity conditioning, 80-100%; reduced intensity conditioning, 60-100%.
* Vital organ function: a) Cardiac: Left ventricular ejection fraction must be > 45% assessed by multigated acquisition (MUGA) scan or echocardiogram. No myocardial infarction within 6 months of transplant evaluation. b) Pulmonary: forced expiratory volume at one second (FEV1), forced vital capacity (FVC), and adjusted diffusing capacity of the lungs for carbon monoxide (DLCO) must be ≥ 50% of predicted values. c) Liver: Transaminases (AST, ALT) less than 2 times upper limit of normal values. d) Kidney: Estimated creatinine clearance ≥ 50 cc/min.
* Signed informed consent.
* Included disease conditions and remission status: a) Acute leukemia in First Complete Remission (CR1) or second/subsequent CR. b) Chronic myeloid leukemia, primary myelofibrosis, chronic myelomonocytic leukemia. c) Int-2 or high risk myelodysplastic syndrome (MDS). d) Hodgkin lymphoma beyond CR1 with chemosensitive disease, Stable Disease (SD) may be included if no mass >3 cm. e) Non-Hodgkin lymphoma in high risk CR1 or subsequent CR (by clinical, cytogenetic or molecular criteria), primary induction failure (PIF) or relapsed with chemosensitive disease. SD may be included if no mass >3 cm. f) Multiple myeloma in CR/Very Good Partial Response (VGPR).

Donor Participants:

* Per Moffitt Cancer Center (MCC) Blood and Marrow Transplant (BMT) program practices, an allele level matched (8/8 HLA A, B, C and DR) sibling or unrelated donor is preferred. If a matched donor is not found, mismatched unrelated or haploidentical donors may be considered.
* If a haploidentical donor is considered, parents, children, full siblings and in selected cases, extended family, will have high resolution typing at the MCC HLA laboratory. A familiar haploidentical donor is chosen among those who share at least one HLA-A, B, C, DRB1 and DQB1 haplotype with the patient.
* Patient will be screened for antibodies targeting mismatched HLA antigens in potential haploidentical donors (donor specific antibodies, DSA). Antibody screen and confirmatory testing using Luminex single antigen-bead test will be done.
* Among several potential donors, will choose in order of priority: a) Matched cytomegalovirus (CMV) immunoglobulin G (IgG) serologic status between donor and recipient. b) ABO blood group system-matched donor preferred, then minor ABO mismatch, then major ABO mismatch. c) Younger donor preferred: child, then sibling, and then parent. d) For male recipient, male donor will be preferred. Avoid mother as a donor unless no other choices.

Exclusion Criteria:

Patient Participants:

* Uncontrolled active bacterial, viral, fungal infection.
* Prior allogeneic HCT.
* Unwilling to comply with study requirements.
* Active, progressive or advanced disease based on diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelli Bejanyan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Bejanyan N, Pidala JA, Wang X, Thapa R, Nishihori T, Elmariah H, Lazaryan A, Khimani F, Davila ML, Mishra A, Faramand R, Jain MD, Ochoa L, Perez LE, Liu H, Alsina M, Kharfan-Dabaja MA, Fernandez H, Nieder ML, Locke FL, Anasetti C, Ayala E. A phase 2 trial of GVHD prophylaxis with PTCy, sirolimus, and MMF after peripheral blood haploidentical transplantation. Blood Adv. 2021 Mar 9;5(5):1154-1163. doi: 10.1182/bloodadvances.2020003779. PMID 33635333
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Conditioning/HCT/GVHD Prophylaxis: Pre-HCT Conditioning, HCT, GVHD Prophylaxis.
Period: Overall Study
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 49.5 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade II-IV Acute Graft vs. Host Disease (GVHD)
Description: Cumulative incidence of grade II-IV acute GVHD by day 100 after HCT. Acute GVHD organ staging and assessment of overall grade will use standard consensus criteria. The cumulative incidence of acute and chronic GVHD will be estimated, considering malignancy relapse and non-relapse death as competing risk events.
Time Frame: 100 days post hematopoietic cell transplant (HCT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Number analyzed (Participants) | 32
percentage of participants | 18.8 [7.5 to 34.0]

2. Secondary Outcome: Incidence of Chronic GVHD
Description: Cumulative incidence of chronic GVHD by 1 year. Chronic GVHD diagnosis follow National Institutes of Health (NIH) Consensus guidelines.
Time Frame: 1 year post HCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Number analyzed (Participants) | 32
percentage of participants | 20.0 [7.9 to 36.0]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from transplant to death or last follow-up, and is reported as percentage of surviving participants.
Time Frame: Up to 1 year post HCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Number analyzed (Participants) | 32
percentage of participants | 70.2 [55.5 to 88.6]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival defined by the time interval from transplant to relapse/recurrence, to death or to last follow-up. Reported as percentage of participants who are disease free one year post HCT.
Time Frame: Up to 1 year post HCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
Number analyzed (Participants) | 32
percentage of participants | 56.6 [41.3 to 77.7]

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Arm/Group | Conditioning/HCT/GVHD Prophylaxis
All-Cause Mortality (participants affected / at risk) | 5/32
Serious Adverse Events (participants affected / at risk) | 17/32
Other Adverse Events (participants affected / at risk) | 5/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conditioning/HCT/GVHD Prophylaxis (N=32)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders -Other (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Renal and urinary disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations -Other (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conditioning/HCT/GVHD Prophylaxis (N=32)
Infections and Infestations - Other (Infections and infestations) | 1 (1)
Fever (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03018223/Prot_SAP_000.pdf